CLINICAL TRIAL: NCT00968708
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Cardiovascular Outcomes Following Treatment With Alogliptin in Addition to Standard of Care in Subjects With Type 2 Diabetes and Acute Coronary Syndrome
Brief Title: Cardiovascular Outcomes Study of Alogliptin in Patients With Type 2 Diabetes and Acute Coronary Syndrome
Acronym: EXAMINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-322_402; U1111-1111-6825 (Registry Identifier: WHO); 2009-011222-34 (Registry Identifier: EudraCT); JapicCTI-101246 (Registry Identifier: JapicCTI); DOH-27-0310-3047 (Registry Identifier: SANCTR); 09/H0709/63 (Registry Identifier: NRES); CTRI/2010/091/000046 (Registry Identifier: CTRI); 2009-011222-34 (Registry Identifier: REPEC); 2009-011222-34 (Registry Identifier: OsSC); NMRR-09-872-4471 (Registry Identifier: NMRR)
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Results first posted 2014-04-15 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes Mellitus, Type 2; Acute Coronary Syndrome
Keywords: Diabetes Mellitus - Type 2; Diabetes Mellitus; cardiovascular outcomes; heart attack; stroke; dipeptidyl-peptidase IV inhibitors; metabolic disorders; metabolic diseases; glucose metabolism disorders
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Acute Coronary Syndrome; Diabetes Mellitus; Myocardial Infarction; Stroke; Metabolic Diseases; Glucose Metabolism Disorders | interventions — alogliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Experimental): Alogliptin placebo matching tablets, orally, once daily. Participants continued to receive standard of care for cardiovascular disease and diabetes according to regional guidelines.
  Interventions: Drug: Placebo
- Alogliptin (Experimental): Alogliptin 25 mg, tablets, orally, once daily for participants with normal or mildly impaired renal function as defined by estimated glomerular filtration rate (eGFR) ≥ 60 mL/min). Alogliptin 12.5 mg, tablets, orally, once daily for participants with moderately impaired renal function (eGFR ≥30 and <60 mL/min). Alogliptin 6.25 mg, tablets, orally, once daily for participants with severely impaired renal function or end stage renal disease (eGFR <30 mL/min). Participants continued to receive standard of care for cardiovascular disease and diabetes according to regional guidelines.
  Interventions: Drug: Alogliptin

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets
  Other Names: Nesina®; SYR-322; SYR110322
  Arms: Alogliptin
Drug: Placebo — Alogliptin placebo matching tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the cardiovascular outcomes of alogliptin, once daily (QD), compared with placebo, in addition to standard of care, in patients with type 2 diabetes mellitus and acute coronary syndrome.

DETAILED DESCRIPTION:
Alogliptin is a selective and potent dipeptidyl peptidase-4 inhibitor developed by Takeda for use in patients with type 2 diabetes mellitus.

Cardiovascular outcomes is of special interest in the type 2 diabetes mellitus population, particularly in type 2 diabetes mellitus patients who have cardiovascular disease and are at high risk for major adverse cardiac events, such as those patients who have had recent acute coronary syndrome.

This study has been designed to evaluate the cardiovascular safety of alogliptin versus placebo in addition to Standard of Care in adults with type 2 diabetes mellitus and acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus
* Is receiving monotherapy or combination antidiabetic therapy with a glycosylated hemoglobin level between 6.5% and 11.0%, inclusive, at Screening (between 7.0 and 11.0%, inclusive, if the participant's antidiabetic regimen includes insulin)
* Diagnosis of acute coronary syndrome within 15 to 90 days prior to randomization.

Exclusion Criteria:

* Signs of type 1 diabetes mellitus
* Currently receiving a glucagon-like peptide-1 analogue for glycemic control of type 2 diabetes mellitus at Screening
* Received a dipeptidyl peptidase-4 inhibitor for either more than 14 days total or within the 3 months prior to Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5380 (Actual)
Dates: Start 2009-09; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (908):
- United States (292):
  - Birmingham, Alabama
  - Dothan, Alabama
  - Mobile, Alabama
  - Muscle Shoals, Alabama
  - Cottonwood, Arizona
  - Goodyear, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Malvern, Arkansas
  - Searcy, Arkansas
  - White Hall, Arkansas
  - Alameda, California
  - Aliso Viejo, California
  - Anaheim, California
  - Bell Gardens, California
  - Beverly Hills, California
  - Chula Vista, California
  - Corona, California
  - Downey, California
  - Escondido, California
  - Fullerton, California
  - Huntington Beach, California
  - Huntington Park, California
  - Inglewood, California
  - La Mirada, California
  - Lakewood, California
  - Lancaster, California
  - Lomita, California
  - Long Beach, California
  - Los Angeles, California
  - Los Gatos, California
  - Merced, California
  - Newport Beach, California
  - Northridge, California
  - Oakland, California
  - Palm Springs, California
  - Pomona, California
  - San Diego, California
  - San Dimas, California
  - Santa Ana, California
  - Santa Clarita, California
  - Stockton, California
  - Tarzana, California
  - Torrence, California
  - Van Nuys, California
  - Ventura, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Bridgeport, Connecticut
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Brandon, Florida
  - Davie, Florida
  - Daytona Beach, Florida
  - Delray Beach, Florida
  - Doral, Florida
  - Fleming Island, Florida
  - Fort Lauderdale, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Lake Mary, Florida
  - Largo, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Miami Lakes, Florida
  - Naples, Florida
  - New Smyrna Beach, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Panama City, Florida
  - Pembroke Pines, Florida
  - Pensacola, Florida
  - Saint Cloud, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Stuart, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Cartersville, Georgia
  - Conyers, Georgia
  - Dunwoody, Georgia
  - Marietta, Georgia
  - Savannah, Georgia
  - Tucker, Georgia
  - Waycross, Georgia
  - Nampa, Idaho
  - Aurora, Illinois
  - Boilingbrook, Illinois
  - Bolingbrook, Illinois
  - Burr Ridge, Illinois
  - Chicago, Illinois
  - Jerseyville, Illinois
  - Melrose Park, Illinois
  - Moline, Illinois
  - Peoria, Illinois
  - Quincy, Illinois
  - Springfield, Illinois
  - Elkhart, Indiana
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Muncie, Indiana
  - Munster, Indiana
  - New Albany, Indiana
  - Valparaiso, Indiana
  - Council Bluffs, Iowa
  - Shawnee Mission, Kansas
  - Elizabethtown, Kentucky
  - Lexington, Kentucky
  - Madisonville, Kentucky
  - Owensboro, Kentucky
  - Alexandria, Louisiana
  - Houma, Louisiana
  - Lafayette, Louisiana
  - Natchitoches, Louisiana
  - New Orleans, Louisiana
  - Slidell, Louisiana
  - Biddeford, Maine
  - Rockport, Maine
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Oxon Hill, Maryland
  - Rockville, Maryland
  - Boston, Massachusetts
  - Brockton, Massachusetts
  - Fall River, Massachusetts
  - Alpena, Michigan
  - Bridgman, Michigan
  - Dearborn, Michigan
  - Detroit, Michigan
  - Kalamazoo, Michigan
  - Lapeer, Michigan
  - Livonia, Michigan
  - Midland, Michigan
  - Muskegon, Michigan
  - Saginaw, Michigan
  - Troy, Michigan
  - Warren, Michigan
  - Waterford, Michigan
  - Ypsilanti, Michigan
  - Duluth, Minnesota
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Chesterfield, Missouri
  - Jefferson City, Missouri
  - Kansas City, Missouri
  - Saint Joseph, Missouri
  - St Louis, Missouri
  - Great Falls, Montana
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Pahrump, Nevada
  - Brick, New Jersey
  - Bridgewater, New Jersey
  - Camden, New Jersey
  - Fort Lee, New Jersey
  - Haddon Heights, New Jersey
  - Linden, New Jersey
  - New Brunswick, New Jersey
  - Newark, New Jersey
  - Ridgewood, New Jersey
  - Sewell, New Jersey
  - Sicklerville, New Jersey
  - South Plainfield, New Jersey
  - Albuquerque, New Mexico
  - Cortlandt Manor, New York
  - Freeport, New York
  - Huntington, New York
  - Johnson City, New York
  - Kingston, New York
  - New Hartford, New York
  - New York, New York
  - Rochester, New York
  - Saratoga Springs, New York
  - Springfield Gardens, New York
  - The Bronx, New York
  - Valhalla, New York
  - Williamsville, New York
  - Asheville, North Carolina
  - Burlington, North Carolina
  - Charlotte, North Carolina
  - Elizabeth City, North Carolina
  - Forsyth, North Carolina
  - Greensboro, North Carolina
  - Hickory, North Carolina
  - Lenoir, North Carolina
  - Smithfield, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Minot, North Dakota
  - Akron, Ohio
  - Athens, Ohio
  - Berea, Ohio
  - Boardman, Ohio
  - Carlisle, Ohio
  - Centerville, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Franklin, Ohio
  - Lorain, Ohio
  - Marion, Ohio
  - Maumee, Ohio
  - Middleburg Heights, Ohio
  - Springfield, Ohio
  - Toledo, Ohio
  - Westlake, Ohio
  - Zanesville, Ohio
  - Bartlesville, Oklahoma
  - Oklahoma City, Oklahoma
  - Yukon, Oklahoma
  - Bend, Oregon
  - Corvallis, Oregon
  - Hillsboro, Oregon
  - Portland, Oregon
  - Altoona, Pennsylvania
  - Bethlehem, Pennsylvania
  - Clymer, Pennsylvania
  - Fleetwood, Pennsylvania
  - Langhorne, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Schwenksville, Pennsylvania
  - Scotland, Pennsylvania
  - Sellersville, Pennsylvania
  - Yardley, Pennsylvania
  - East Providence, Rhode Island
  - Beaufort, South Carolina
  - Easley, South Carolina
  - Florence, South Carolina
  - Spartanburg, South Carolina
  - Taylors, South Carolina
  - Sioux Falls, South Dakota
  - Bartlett, Tennessee
  - Bristol, Tennessee
  - Cleveland, Tennessee
  - Franklin, Tennessee
  - Germantown, Tennessee
  - Jackson, Tennessee
  - Johnson City, Tennessee
  - Kingsport, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Murfreesboro, Tennessee
  - Nashville, Tennessee
  - Oak Ridge, Tennessee
  - Austin, Texas
  - Beaumont, Texas
  - Carrollton, Texas
  - Dallas, Texas
  - Denton, Texas
  - Edinburg, Texas
  - Fort Worth, Texas
  - Grapevine, Texas
  - Houston, Texas
  - McKinney, Texas
  - North Richland Hills, Texas
  - Plano, Texas
  - Saginaw, Texas
  - San Antonio, Texas
  - Southlake, Texas
  - Temple, Texas
  - Tomball, Texas
  - Bountiful, Utah
  - Ogden, Utah
  - Salt Lake City, Utah
  - Bennington, Vermont
  - South Burlington, Vermont
  - Burke, Virginia
  - Charlottesville, Virginia
  - Galax, Virginia
  - Lakeridge, Virginia
  - Manassas, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Roanoke, Virginia
  - Suffolk, Virginia
  - Virginia Beach, Virginia
  - Everett, Washington
  - Tacoma, Washington
  - Beloit, Wisconsin
  - Green Bay, Wisconsin
  - Madison, Wisconsin
  - Manitowoc, Wisconsin
  - Milwaukee, Wisconsin
  - Waukesha, Wisconsin
- Argentina (37):
  - Bahía Blanca
  - Buenos Aires
  - C0rdoba
  - Capital Federal, Buenos Aires
  - Capital Federal
  - Carlos Paz, C0rdoba
  - Ciudad Aut0noma de Buenos Aires
  - Ciudad de C0rdoba
  - Cordoba - Cordoba
  - Corrientes
  - Córdoba
  - Derqui Pilar, Buenos Aires
  - Formosa
  - Haedo, Buenos Aires
  - La Plata
  - La Plata, Buenos Aires
  - Mar del Plata
  - Mar Del Plata, Provincia de Buenos Aires
  - Mendoza
  - Moron, Buenos Aires
  - Olivos
  - Quilmes
  - Ramos Mejia, Buenos Aries
  - Ramos Mejía
  - Rosario
  - Rosario - Santa Fe
  - Rosario, Provincia de Santa Fe
  - Salta
  - San Isidro
  - San Juan, San Juan
  - San Justo
  - San Luis
  - San Miguel de Tucumán
  - San Salvador de Jujuy
  - Santa Fe
  - Trelew, Chubut
  - Villa María
- Australia (11):
  - Broken Hill, New South Wales
  - Kogarah, New South Wales
  - Milton, Queensland
  - Nambour, Queensland
  - Hobart, Tasmania
  - Fitzroy, Victoria
  - Frankston, Victoria
  - Heidelberg, Victoria
  - Prahran, Victoria
  - Adelaide, SA
  - Bruce
- Austria (4):
  - Feldkirch
  - Graz
  - Salzburg
  - Vienna
- Belgium (6):
  - Antwerp
  - Bonheiden
  - Brasschaat
  - Brussels
  - Ghent
  - La Louvière
- Brazil (50):
  - Curitiba, Paraná
  - Rio de Janeiro, Rio de Janeiro
  - São Paulo, São Paulo
  - Tatuí, São Paulo
  - Aracaju, Sergipe
  - Belem - PA
  - Belo Horizonte - MG
  - Belo Horizonte, Minas Gerais
  - Blumenau
  - Brasilia - DF
  - Brasilia, Distrito Federal
  - Campina Grande do Sul
  - Campinas, Sao Paulo
  - Campo Grande, Mato Grosso Do Sul
  - Curitiba, Parana
  - Fortaleza - CE
  - Fortaleza, Ceara
  - Goiania, Goias
  - Goiânia
  - Joinville
  - Londrina/PR
  - Macei0
  - Marilia, Sao Paulo
  - Marília
  - Mogi das Cruzes
  - Natal
  - Natal, RN
  - Passo Fundo, Rio Grande Do Sul
  - Porto Alegre
  - Porto Alegre - RS
  - Porto Alegre, Rio Grande Do Sul
  - Recife
  - Recife, PE
  - Recife, Pernambuco
  - Rio de Janeiro
  - Rio de Janeiro - RJ
  - Salvador - BA
  - Salvador, Bahia
  - Santo André
  - Sao Jose Do Rio Preto, Sao Paulo
  - Sao Jose Do Rio Preto- SP
  - Sao Jose, Santa Catarina
  - Sao Paulo, Sao Paulo
  - Sao Paulo, SP
  - São José do Rio Preto
  - São Paulo
  - Sobral, CE
  - Taguatinga
  - Uberlandia, Minas Gerais
  - Votuporanga
- Bulgaria (11):
  - Blagoevgrad
  - Dimitrovgrad
  - Kazanlak
  - Lovech
  - Pleven
  - Plovdiv
  - Sevlievo
  - Smolyan
  - Sofia
  - Stara Zagora
  - Varna
- Canada (30):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Abbotsford, British Columbia
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Grand Falls-Windsor, Newfoundland and Labrador
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Ajax, Ontario
  - Cambridge, Ontario
  - Greater Sudbury, Ontario
  - Hamilton, Ontario
  - Newmarket, Ontario
  - Niagara Falls, Ontario
  - Ontario, Ontario
  - Oshawa, Ontario
  - Pickering, Ontario
  - Smiths Falls, Ontario
  - Toronto, Ontario
  - Greenfield Park, Quebec
  - Greenfield, Quebec
  - Lachine, Quebec
  - Mount Royal, Quebec
  - Pointe-Claire, Quebec
  - Québec, Quebec
  - Saint-Jérôme, Quebec
  - Sainte-Foy, Quebec
  - Sherbrooke, Quebec
  - Terrebonne, Quebec
- Chile (10):
  - Antofagasta
  - Antofagasta, Region II
  - Iquique, Region I
  - Osorno
  - Rancagua
  - Santiago
  - Talcahuano
  - Temuco
  - Temuco, Region de La Araucania
  - Viña del Mar
- Colombia (4):
  - Barranquilla
  - Bogotá
  - Bucaramanga
  - Medellín
- Croatia (9):
  - Čakovec
  - Krapinske Toplice
  - Osijek
  - Rijeka
  - Sisak
  - Split
  - Virovitica
  - Zadar
  - Zagreb
- Czechia (6):
  - Čáslav
  - Hradec Králové
  - Olomouc
  - Ostrava - Vitkovice
  - Zlín
  - Znojmo
- Denmark (3):
  - Herlev
  - Herning
  - København NV
- Egypt (3):
  - Alexandria
  - Giza
  - Monofia
- Finland (6):
  - Helsinki
  - Jyväskylä
  - Kokkola
  - Kuopio
  - Tampere
  - Turku
- France (13):
  - Bordeaux
  - Corbeil-Essonnes
  - Créteil
  - Dijon
  - La Rochelle
  - Lille
  - Montpellier
  - Narbonne
  - Paris
  - Pau
  - Pessac
  - Rennes
  - Toulouse
- Germany (20):
  - Bad Nauheim
  - Bensheim
  - Berlin
  - Cologne
  - Dortmund
  - Dresden
  - Essen
  - Halle
  - Jena
  - Kassel
  - Leipzig
  - Mainz
  - Mannheim
  - München
  - Münster
  - Neumünster
  - Neuwied
  - Sankt Ingbert
  - Siegen
  - Wangen
- Marousi, Greece
- Guatemala (2):
  - Guatemala City
  - Quetzaltenango
- Hong Kong (4):
  - Hong Kong
  - Kowloon
  - Shatin
  - Tsuen Wan
- Hungary (15):
  - Budaörs
  - Budapest
  - Debrecen
  - Dunaújváros
  - Gyula
  - H0dmezovasarhely
  - Kaposvár
  - Kecskemét
  - Nagykanizsa
  - Pécs
  - Sopron
  - Szentes
  - Székesfehérvár
  - Szombathely
  - Zalaegerszeg
- India (32):
  - Hyderabad, Andhra Pradesh
  - Nellore, Andhra Pradesh
  - Vijayawada, Andhra Pradesh
  - Visakhapatnam, Andhra Pradesh
  - Perumbākkam, Chennai
  - Ahmedabad, Gujarat
  - Anand, Gujarat
  - Surat, Gujarat
  - Vadodara, Gujarat
  - Bangalore, Karnataka
  - Belagavi, Karnataka
  - Mangalore, Karnataka
  - Manipal, Karnataka
  - Mysore, Karnataka
  - Kochi, Kerala
  - Thiruvananthapuram, Kerala
  - Thrissur, Kerala
  - Trivandrum, Kerala
  - Aurangabad, Maharashtra
  - Mumbai, Maharashtra
  - Nagpur, Maharashtra
  - Nashik, Maharashtra
  - Pune, Maharashtra
  - Delhi, National Capital Territory of Delhi
  - New Delhi, National Capital Territory of Delhi
  - Jalandhar, Punjab
  - Ludhiana, Punjab
  - Jaipur, Rajasthan
  - Chennai, Tamil Nadu
  - Coimbatore, Tamil Nadu
  - Madurai, Tamil Nadu
  - Kolkata, West Bengal
- Israel (14):
  - Ashkelon
  - Beersheba
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Nahariya
  - Nazareth
  - Petah Tikva
  - Rehovot
  - Rishon LeZiyyon
  - Safed
  - Tel Aviv
  - Tiberias
- Italy (9):
  - Cosenza
  - Isernia
  - Milan
  - Napoli
  - Palermo
  - Pavia
  - Ravenna
  - Roma
  - Sesto San Giovanni
- Japan (45):
  - Aichi-gun, Aichi-ken
  - Nagoya, Aichi-ken
  - Seto, Aichi-ken
  - Funabashi, Chiba
  - Kashiwa, Chiba
  - Imabari, Ehime
  - Fukuoka, Fukuoka
  - Kasuga, Fukuoka
  - Kitakyushu, Fukuoka
  - Ohkawa-city, Fukuoka
  - Fukushima, Fukushima
  - Gifu, Gifu
  - Shibukawa, Gunma
  - Takasaki, Gunma
  - Higashihiroshima, Hiroshima
  - Tomakomai, Hokkaido
  - Amagasaki, Hyōgo
  - Kanazawa, Ishikawa-ken
  - Sakaidechō, Kagawa-ken
  - Kawasaki, Kanagawa
  - Sagamihara-shi, Kanagawa
  - Nankoku, Kochi
  - Kumamoto, Kumamoto
  - Uji-shi, Kyoto
  - Matsusaka, Mie-ken
  - Nagasaki, Nagasaki
  - Niigata, Niigata
  - Ōita, Oita Prefecture
  - Okayama, Okayama-ken
  - Shimajiri-gun, Okinawa
  - Tomigusuku, Okinawa
  - Kishiwada, Osaka
  - Matsubara, Osaka
  - Yao-shi, Osaka
  - Saga, Saga-ken
  - Ageo, Saitama
  - Wako, Saitama
  - Hamada, Shimane
  - Suntou-gun, Shizuoka
  - Komatsushimachō, Tokushima
  - Tokushima, Tokushima
  - Hino, Tokyo
  - Tachikawa, Tokyo
  - Tokyo, Tokyo
  - Iwakuni-shi, Yamaguchi
- Dasman, Kuwait
- Latvia (5):
  - Daugavpils
  - Ogre
  - Riga
  - Tukums
  - Valmiera
- Lithuania (6):
  - Kaunas
  - Kėdainiai
  - Klaipėda
  - Palanga
  - Panevezys
  - Vilnius
- Malaysia (8):
  - Alor Star
  - Batu Caves
  - George Town
  - Kuala Lumpur
  - Kuala Selangor
  - Kuantan
  - Kubang Kerian
  - Pulau Pinang
- Mexico (33):
  - Acapulco, Guerrero
  - Aguascalientes
  - Chihuahua City
  - Chihuhua, Chihuhua
  - Ciudad Obregon, Sonora
  - Cuernavaca
  - Cuernavaca, Morelos
  - Culiacán
  - Durango
  - Guadalajara
  - Guadalajara, Jalisco
  - Merida, Yucatan
  - Metepec
  - Mexicali, Baja California
  - Mexico City
  - Mexico City, Mexico
  - México
  - Monclova, Coahuila
  - Monterrey
  - Monterrey, NL
  - Monterrey, Nuevo Le0n
  - Monterrey, Nuevo Leon
  - Morelia, Michoacan
  - Pachuca
  - Saltillo
  - Saltillo, Coahuila
  - San Luis Potosi.SLP
  - San Luis Potosí City
  - Tijuana, Baja California Norte
  - Tlalnepantla
  - Tlalnepantla, Edo de Mexico
  - Xalapa, Veracruz
  - Zapopan
- New Zealand (6):
  - Auckland
  - Christchurch
  - Otahuhu
  - Palmerston North
  - Takapuna
  - Tauranga
- Peru (16):
  - Arequipa
  - Bellavista
  - Callao
  - Cusco
  - Huacho
  - Ica
  - La Victoria, Lima
  - Lima
  - Lima San Isidro
  - Los Olivos
  - Miraflores, Lima
  - Piura
  - San Isidro, Lima
  - San Miguel, Lima
  - Trujillo
  - Trujillo, La Libertad
- Philippines (10):
  - Baguio City
  - Dasmariñas
  - Davao City
  - Iloilo City
  - Laoag
  - Makati City
  - Manila
  - Marikina City
  - Pasig
  - Quezon City
- Poland (28):
  - Bialystok
  - Bydgoszcz
  - Częstochowa
  - Dąbrowa Górnicza
  - Elblag
  - Gdansk
  - Gdynia
  - Grodzisk Mazowiecki
  - Inowrocław
  - Katowice
  - Kielce
  - Krakow
  - Legnica
  - Lodz
  - Lubartów
  - Lublin
  - Puławy
  - Płock
  - Radom
  - Ruda Śląska
  - Skierniewice
  - Szczecin
  - Słupsk
  - Torun
  - Warsaw
  - Wroclaw
  - Zabrze
  - Zgierz
- Portugal (4):
  - Coimbra
  - Faro
  - Lisbon
  - Vila Real
- Puerto Rico (11):
  - Aibonito, PR
  - Halo Rey, PR
  - Ponce, PR
  - Salinas, PR
  - Santurce, PR
  - Carolina
  - Cidra
  - Levittown
  - Manatí
  - Mayagüez
  - San Juan
- Romania (13):
  - Bacau
  - Baia Mare
  - Brasov
  - Brăila
  - Bucharest
  - Buzău
  - Galati
  - Iași
  - Oradea
  - Ploieşti
  - Satu Mare
  - Târgu Mureş
  - Timișoara
- Russia (17):
  - Arkhangelsk
  - Barnaul
  - Ivanovo
  - Kazan'
  - Kemerovo
  - Krasnodar
  - Krasnoyarsk
  - Kursk
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Rostov-on-Don
  - Saint Petersburg
  - Saratov
  - Ufa
  - Volgograd
  - Vsevolozhsk
- Serbia (2):
  - Belgrade
  - Niš
- Slovakia (15):
  - Bardejov
  - Bratislava
  - Dolný Kubín
  - Komárno
  - Kosice - Saca
  - Košice
  - Levice
  - Liptovský Hrádok
  - Nové Mesto nad Váhom
  - Nové Zámky
  - Považská Bystrica
  - Rimavská Sobota
  - Ružomberok
  - Svidník
  - Žilina
- South Africa (11):
  - Port Elizabeth, Eastern Cape
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - Durban, KwaZulu-Natal
  - Cape Town, Western Cape
  - Paarl, Western Cape
  - Somerset West, Western Cape
  - Tygerberg, Western Cape
  - Worcester, Western Cape
  - Durban
  - Pretoria
- South Korea (12):
  - Anyang
  - Busan
  - Daegu
  - Goyang-si
  - Guri-si
  - Gyeonggi-do
  - Jeonju
  - Kangwon-do
  - Pusan
  - Seoul
  - Suwon
  - Yangsan
- Spain (11):
  - Zaragoza, Arag0n
  - Cuenca, Castille-La Mancha
  - Barcelona, Catalonia
  - Figueres, Catalonia
  - A Coruña, Galicia
  - Santiago de Compostela, Galicia
  - Oviedo, Principality of Asturias
  - Torrevieja, Valencia
  - Bacarot
  - Mérida
  - Palma de Mallorca
- Sweden (8):
  - Dalby
  - Falköping
  - Gothenburg
  - Härnösand
  - Kristianstad
  - Malmo
  - Motala
  - Stockholm
- Taiwan (3):
  - Kaohsiung City
  - Taipei County
  - Taoyuan District
- Thailand (11):
  - Amphure Muang
  - Bangkojk
  - Bangkok
  - Chiang Mai
  - Chiang Rai
  - Muang
  - Nakhon Ratchasima
  - Pathumwan
  - Patumthani
  - Phitsanulok
  - Phrae
- Turkey (Türkiye) (5):
  - Ankara, Balgat
  - Antalya
  - Istanbul
  - Kayseri
  - Konya
- Ukraine (10):
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kyiv
  - Lviv
  - Odesa
  - Poltava
  - Simferopol
  - Vinnytsia
  - Zaporizhzhya
- Abu Dhabi, United Arab Emirates
- United Kingdom (24):
  - Barnsley
  - Bath
  - Birmingham
  - Bournemouth
  - Carshalton
  - Chertsey
  - Chichester
  - Colchester
  - Coventry
  - Croydon
  - Doncaster
  - Glasgow
  - Hull
  - Inverness
  - Kirkcaldy
  - Liverpool
  - Livingston
  - London
  - Nuneaton
  - Stevenage
  - Sunderland
  - Torquay
  - Wakefield
  - West Midlands

REFERENCES:
- [Derived] Ferreira JP, Rossignol P, Bakris G, Mehta C, White WB, Zannad F. Blood and Urine Biomarkers Predicting Worsening Kidney Function in Patients with Type 2 Diabetes Post-Acute Coronary Syndrome: An Analysis from the EXAMINE Trial. Am J Nephrol. 2021;52(12):969-976. doi: 10.1159/000519436. Epub 2021 Dec 6. PMID 34872085
- [Derived] Ferreira JP, Mehta C, Sharma A, Nissen SE, Rossignol P, Zannad F. Alogliptin after acute coronary syndrome in patients with type 2 diabetes: a renal function stratified analysis of the EXAMINE trial. BMC Med. 2020 Jun 4;18(1):165. doi: 10.1186/s12916-020-01616-8. PMID 32493335
- [Derived] Sharma A, Vaduganathan M, Ferreira JP, Liu Y, Bakris GL, Cannon CP, White WB, Zannad F. Clinical and Biomarker Predictors of Expanded Heart Failure Outcomes in Patients With Type 2 Diabetes Mellitus After a Recent Acute Coronary Syndrome: Insights From the EXAMINE Trial. J Am Heart Assoc. 2020 Jan 7;9(1):e012797. doi: 10.1161/JAHA.119.012797. Epub 2020 Jan 4. PMID 31902327
- [Derived] White WB, Jalil F, Cushman WC, Bakris GL, Bergenstal R, Heller SR, Liu Y, Mehta C, Zannad F, Cannon CP. Average Clinician-Measured Blood Pressures and Cardiovascular Outcomes in Patients With Type 2 Diabetes Mellitus and Ischemic Heart Disease in the EXAMINE Trial. J Am Heart Assoc. 2018 Oct 16;7(20):e009114. doi: 10.1161/JAHA.118.009114. PMID 30371278
- [Derived] Jarolim P, White WB, Cannon CP, Gao Q, Morrow DA. Serial Measurement of Natriuretic Peptides and Cardiovascular Outcomes in Patients With Type 2 Diabetes in the EXAMINE Trial. Diabetes Care. 2018 Jul;41(7):1510-1515. doi: 10.2337/dc18-0109. Epub 2018 May 30. PMID 29848776
- [Derived] Sharma A, Cannon CP, White WB, Liu Y, Bakris GL, Cushman WC, Zannad F. Early and Chronic Dipeptidyl-Peptidase-IV Inhibition and Cardiovascular Events in Patients With Type 2 Diabetes Mellitus After an Acute Coronary Syndrome: A Landmark Analysis of the EXAMINE Trial. J Am Heart Assoc. 2018 May 16;7(11):e007649. doi: 10.1161/JAHA.117.007649. PMID 29769203
- [Derived] White WB, Heller SR, Cannon CP, Howitt H, Khunti K, Bergenstal RM; EXAMINE Investigators. Alogliptin in Patients with Type 2 Diabetes Receiving Metformin and Sulfonylurea Therapies in the EXAMINE Trial. Am J Med. 2018 Jul;131(7):813-819.e5. doi: 10.1016/j.amjmed.2018.02.023. Epub 2018 Mar 23. PMID 29581078
- [Derived] Hwang YC, Morrow DA, Cannon CP, Liu Y, Bergenstal R, Heller S, Mehta C, Cushman W, Bakris GL, Zannad F, White WB. High-sensitivity C-reactive protein, low-density lipoprotein cholesterol and cardiovascular outcomes in patients with type 2 diabetes in the EXAMINE (Examination of Cardiovascular Outcomes with Alogliptin versus Standard of Care) trial. Diabetes Obes Metab. 2018 Mar;20(3):654-659. doi: 10.1111/dom.13136. Epub 2017 Nov 21. PMID 29064626
- [Derived] Kay S, Strickson A, Puelles J, Selby R, Benson E, Tolley K. Comparative Effectiveness of Adding Alogliptin to Metformin Plus Sulfonylurea with Other DPP-4 Inhibitors in Type 2 Diabetes: A Systematic Review and Network Meta-Analysis. Diabetes Ther. 2017 Apr;8(2):251-273. doi: 10.1007/s13300-017-0245-8. Epub 2017 Mar 8. PMID 28275958
- [Derived] Cavender MA, White WB, Jarolim P, Bakris GL, Cushman WC, Kupfer S, Gao Q, Mehta CR, Zannad F, Cannon CP, Morrow DA. Serial Measurement of High-Sensitivity Troponin I and Cardiovascular Outcomes in Patients With Type 2 Diabetes Mellitus in the EXAMINE Trial (Examination of Cardiovascular Outcomes With Alogliptin Versus Standard of Care). Circulation. 2017 May 16;135(20):1911-1921. doi: 10.1161/CIRCULATIONAHA.116.024632. Epub 2017 Feb 28. PMID 28246236
- [Derived] White WB, Kupfer S, Zannad F, Mehta CR, Wilson CA, Lei L, Bakris GL, Nissen SE, Cushman WC, Heller SR, Bergenstal RM, Fleck PR, Cannon CP; EXAMINE Investigators. Cardiovascular Mortality in Patients With Type 2 Diabetes and Recent Acute Coronary Syndromes From the EXAMINE Trial. Diabetes Care. 2016 Jul;39(7):1267-73. doi: 10.2337/dc16-0303. Epub 2016 Jun 11. PMID 27289121
- [Derived] Zannad F, Cannon CP, Cushman WC, Bakris GL, Menon V, Perez AT, Fleck PR, Mehta CR, Kupfer S, Wilson C, Lam H, White WB; EXAMINE Investigators. Heart failure and mortality outcomes in patients with type 2 diabetes taking alogliptin versus placebo in EXAMINE: a multicentre, randomised, double-blind trial. Lancet. 2015 May 23;385(9982):2067-76. doi: 10.1016/S0140-6736(14)62225-X. Epub 2015 Mar 10. PMID 25765696
- [Derived] White WB, Cannon CP, Heller SR, Nissen SE, Bergenstal RM, Bakris GL, Perez AT, Fleck PR, Mehta CR, Kupfer S, Wilson C, Cushman WC, Zannad F; EXAMINE Investigators. Alogliptin after acute coronary syndrome in patients with type 2 diabetes. N Engl J Med. 2013 Oct 3;369(14):1327-35. doi: 10.1056/NEJMoa1305889. Epub 2013 Sep 2. PMID 23992602
- [Derived] White WB, Bakris GL, Bergenstal RM, Cannon CP, Cushman WC, Fleck P, Heller S, Mehta C, Nissen SE, Perez A, Wilson C, Zannad F. EXamination of cArdiovascular outcoMes with alogliptIN versus standard of carE in patients with type 2 diabetes mellitus and acute coronary syndrome (EXAMINE): a cardiovascular safety study of the dipeptidyl peptidase 4 inhibitor alogliptin in patients with type 2 diabetes with acute coronary syndrome. Am Heart J. 2011 Oct;162(4):620-626.e1. doi: 10.1016/j.ahj.2011.08.004. Epub 2011 Sep 14. PMID 21982652

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 898 investigative sites worldwide from 24 September 2009 to 18 June 2013.
Pre-assignment Details: Participants with a diagnosis of type 2 diabetes mellitus and acute coronary syndrome were enrolled equally in 1 of 2 treatment groups, once a day placebo or alogliptin, in addition to receiving standard of care for cardiovascular disease and diabetes.
Period: Overall Study
Arm/Group | Placebo | Alogliptin
Started | 2679 | 2701
Treated | 2676 | 2698
Completed | 2361 | 2403
Not Completed | 318 | 298
Not completed — Adverse Event | 169 | 150
Not completed — Major Protocol Deviation | 0 | 1
Not completed — Lost to Follow-up | 19 | 11
Not completed — Voluntary Withdrawal | 104 | 101
Not completed — Investigator Discretion | 0 | 1
Not completed — Other | 26 | 34

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) - all randomized participants who signed informed consent.
Groups:
- Placebo: Alogliptin placebo matching tablets, orally, once daily.
- Alogliptin: Alogliptin 25 mg, tablets, orally, once daily for participants with normal or mildly impaired renal function as defined by estimated glomerular filtration rate (eGFR) ≥ 60 mL/min). Alogliptin 12.5 mg, tablets, orally, once daily for participants with moderately impaired renal function (eGFR ≥30 and <60 mL/min). Alogliptin 6.25 mg, tablets, orally, once daily for participants with severely impaired renal function or end stage renal disease (eGFR <30 mL/min).
- Total: Total of all reporting groups
Arm/Group | Placebo | Alogliptin | Total
Number analyzed (Participants) | 2679 | 2701 | 5380
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (9.88) | 61.0 (9.96) | 60.9 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 856 | 873 | 1729
  Male | 1823 | 1828 | 3651
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 54 | 56 | 110
  Asian | 542 | 547 | 1089
  Black or African American | 115 | 101 | 216
  Native Hawaiian or Other Pacific Islander | 5 | 6 | 11
  White | 1943 | 1966 | 3909
  More than one race | 20 | 25 | 45
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 764 | 773 | 1537
  Non-Hispanic or Latino | 1915 | 1928 | 3843
Region of Enrollment [Number; unit: participants]
  Argentina | 136 | 136 | 272
  Australia | 7 | 8 | 15
  Austria | 8 | 8 | 16
  Belgium | 11 | 12 | 23
  Brazil | 179 | 181 | 360
  Bulgaria | 41 | 41 | 82
  Canada | 54 | 55 | 109
  Chile | 51 | 55 | 106
  Colombia | 15 | 13 | 28
  Croatia | 38 | 39 | 77
  Czech Republic | 13 | 13 | 26
  Denmark | 3 | 3 | 6
  Egypt | 7 | 7 | 14
  Finland | 12 | 10 | 22
  France | 11 | 11 | 22
  Germany | 26 | 27 | 53
  Greece | 0 | 1 | 1
  Guatemala | 25 | 24 | 49
  Hong Kong | 11 | 12 | 23
  Hungary | 60 | 59 | 119
  India | 165 | 165 | 330
  Israel | 100 | 101 | 201
  Italy | 25 | 25 | 50
  Japan | 105 | 104 | 209
  Kuwait | 2 | 3 | 5
  Latvia | 6 | 6 | 12
  Lithuania | 16 | 20 | 36
  Malaysia | 39 | 42 | 81
  Mexico | 192 | 191 | 383
  New Zealand | 13 | 13 | 26
  Peru | 79 | 81 | 160
  Philippines | 52 | 50 | 102
  Poland | 121 | 118 | 239
  Portugal | 13 | 16 | 29
  Puerto Rico | 16 | 19 | 35
  Korea, Republic Of | 61 | 62 | 123
  Romania | 40 | 38 | 78
  Russian Federation | 153 | 151 | 304
  Serbia | 35 | 35 | 70
  Slovakia | 46 | 49 | 95
  South Africa | 39 | 41 | 80
  Spain | 21 | 22 | 43
  Sweden | 16 | 16 | 32
  Taiwan, Province Of China | 14 | 13 | 27
  Thailand | 57 | 58 | 115
  Ukraine | 138 | 138 | 276
  United Arab Emirates | 3 | 3 | 6
  United Kingdom | 32 | 34 | 66
  United States | 372 | 372 | 744
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.53 (5.758) | 29.42 (5.422) | 29.48 (5.591)
Duration of Type 2 Diabetes Mellitus [Mean (Standard Deviation); unit: years] | 9.18 (8.121) | 9.13 (8.198) | 9.16 (8.159)
Smoking History [Number; unit: participants]
  Never smoked | 1144 | 1158 | 2302
  Current smoker | 383 | 351 | 734
  Ex-smoker | 1152 | 1192 | 2344
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — Calculated using the Modification of Diet in Renal Disease (MDRD) formula
  mL/min/1.73 m^2 | 71.01 (21.541) | 70.86 (21.297) | 70.93 (21.417)
Renal Impairment Category [Number; unit: participants] — Normal renal function: eGFR ≥90 mL/min/1.73 m^2; Mild renal impairment: eGFR ≥60 and <90 mL/min/1.73 m^2; Moderate renal impairment: eGFR ≥30 and <60 mL/min/1.73 m^2; Severe renal impairment: eGFR <30 mL/min/1.73 m^2; End-stage renal disease (ESRD): eGFR <15 mL/min/1.73 m^2
  participants
    Normal Renal Function | 440 | 399 | 839
    Mild Renal Impairment | 1446 | 1530 | 2976
    Moderate Renal Impairment | 714 | 694 | 1408
    Severe Renal Impairment/End-Stage Renal Disease | 79 | 78 | 157
Index Acute Coronary Syndrome (ACS) Event Type [Number; unit: participants] — Six participants in the placebo arm and 7 participants in the alogliptin arm are not included because they did not meet the ACS requirements for study inclusion.
  participants
    Myocardial Infarction | 2068 | 2084 | 4152
    Unstable Angina | 605 | 609 | 1214
Time From Index ACS Event to Randomization [Mean (Standard Deviation); unit: days] — Six participants in the placebo arm and 7 participants in the alogliptin arm are not included because they did not meet the ACS requirements for study inclusion.
  days | 48.0 (21.95) | 47.6 (22.04) | 47.8 (22.00)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Primary Major Adverse Cardiac Events (MACE)
Description: Primary Major Adverse Cardiac Events were defined as a composite of cardiovascular death, nonfatal myocardial infarction and nonfatal stroke; these events were adjudicated by an independent cardiovascular endpoints committee.
Time Frame: From randomization until the adjudication cut-off date of May 31 2013 (maximum time on study was 41 months).
Population: Full analysis set (all randomized participants)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin
Number analyzed (Participants) | 2679 | 2701
percentage of participants | 11.8 | 11.3
Statistical Analysis 1: Comparison: Placebo vs Alogliptin; Statistical analyses of the primary MACE composite endpoint was based on sequences of 1-sided repeated confidence intervals (CIs) to assess non-inferiority or statistical superiority with respect to the null hypotheses. Each sequence of repeated CIs was constructed using critical values from a 1-sided stopping boundary for a group sequential design (GSD), to preserve an overall false-rejection rate of 2.5%. Each sequence of 1-sided repeated CIs had a simultaneous coverage probability of 97.5%; Test type: Non-Inferiority or Equivalence — If after accrual of 550 participants with MACE events, the upper bound of a 1-sided repeated CI for the hazard ratio (alogliptin to placebo) was <1.0, superiority of alogliptin to placebo for the primary MACE composite would be concluded. If the upper bound of the 1-sided repeated CI for the hazard ratio of the primary MACE composite was <1.3 but ≥1.0 then non-inferiority but not superiority of alogliptin to placebo was to be concluded; p = 0.315, Cox proportional hazards; Hazard Ratio (HR) = 0.962, 97.5% CI 1-sided [upper limit 1.160]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin; Stratified by endpoint renal function and geographic region; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.332, Cox proportional hazards — Stratified by endpoint renal function (defined as the last observed postbaseline renal function (normal renal function/mild renal impairment vs moderate/severe renal impairment including end-stage renal disease)) and geographic region; Hazard Ratio (HR) = 0.965, 97.5% CI 1-sided [upper limit 1.169]

2. Secondary Outcome: Percentage of Participants With Secondary Major Adverse Cardiac Events (MACE)
Description: Secondary MACE composite consisted of cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, or urgent revascularization due to unstable angina; these events were adjudicated by an independent cardiovascular endpoint committee.
Time Frame: From randomization until the adjudication cut-of date of May 31 2013 (maximum time on study was 41 months).
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin
Number analyzed (Participants) | 2679 | 2701
percentage of participants | 13.4 | 12.7
Statistical Analysis 1: Comparison: Placebo vs Alogliptin; Test type: Non-Inferiority or Equivalence — If the upper bound of the confidence interval for the primary MACE composite was <1.0, then statistical superiority of alogliptin to placebo for the secondary MACE composite would be demonstrated; Hazard Ratio (HR) = 0.952, 97.5% CI 1-sided [upper limit 1.135]

ADVERSE EVENTS:
Time Frame: From randomization until the adjudication cut-off date of May 31 2013 (maximum time on study was 41 months).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Alogliptin
Serious Adverse Events (participants affected / at risk) | 952/2679 | 907/2701
Other Adverse Events (participants affected / at risk) | 1493/2679 | 1523/2701
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2679) | Alogliptin (N=2701)
Angina unstable (Cardiac disorders) | 142 | 117
Acute myocardial infarction (Cardiac disorders) | 104 | 125
Angina pectoris (Cardiac disorders) | 83 | 86
Myocardial infarction (Cardiac disorders) | 54 | 66
Cardiac failure congestive (Cardiac disorders) | 53 | 63
Cardiac failure (Cardiac disorders) | 56 | 45
Coronary artery disease (Cardiac disorders) | 34 | 35
Acute coronary syndrome (Cardiac disorders) | 29 | 27
Myocardial ischaemia (Cardiac disorders) | 19 | 20
Atrial fibrillation (Cardiac disorders) | 22 | 15
Coronary artery stenosis (Cardiac disorders) | 17 | 20
Cardiac arrest (Cardiac disorders) | 11 | 14
Cardiogenic shock (Cardiac disorders) | 5 | 14
Cardio-respiratory arrest (Cardiac disorders) | 9 | 6
Ventricular tachycardia (Cardiac disorders) | 10 | 5
Cardiac failure acute (Cardiac disorders) | 8 | 6
Cardiac failure chronic (Cardiac disorders) | 7 | 7
Ischaemic cardiomyopathy (Cardiac disorders) | 4 | 9
Supraventricular tachycardia (Cardiac disorders) | 4 | 7
Ventricular fibrillation (Cardiac disorders) | 6 | 5
Atrial flutter (Cardiac disorders) | 4 | 3
Bradycardia (Cardiac disorders) | 4 | 3
Arrhythmia (Cardiac disorders) | 4 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 6
Cardiomyopathy (Cardiac disorders) | 1 | 4
Left ventricular failure (Cardiac disorders) | 2 | 3
Cardiopulmonary failure (Cardiac disorders) | 1 | 3
Mitral valve incompetence (Cardiac disorders) | 2 | 1
Silent myocardial infarction (Cardiac disorders) | 2 | 1
Tachycardia (Cardiac disorders) | 3 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 1
Atrial tachycardia (Cardiac disorders) | 2 | 0
Cardiac discomfort (Cardiac disorders) | 2 | 0
Cardiorenal syndrome (Cardiac disorders) | 1 | 1
Coronary artery insufficiency (Cardiac disorders) | 0 | 2
Left ventricular dysfunction (Cardiac disorders) | 1 | 1
Postinfarction angina (Cardiac disorders) | 2 | 0
Right ventricular failure (Cardiac disorders) | 1 | 1
Sick sinus syndrome (Cardiac disorders) | 2 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Cardiac asthma (Cardiac disorders) | 1 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Cor pulmonale chronic (Cardiac disorders) | 1 | 0
Coronary artery dissection (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Coronary artery thrombosis (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Nodal rhythm (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Trifascicular block (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricular dysfunction (Cardiac disorders) | 1 | 0
Ventricular dyskinesia (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 44 | 49
Sepsis (Infections and infestations) | 19 | 11
Bronchitis (Infections and infestations) | 10 | 14
Urinary tract infection (Infections and infestations) | 14 | 10
Cellulitis (Infections and infestations) | 15 | 7
Gastroenteritis (Infections and infestations) | 10 | 7
Septic shock (Infections and infestations) | 6 | 10
Postoperative wound infection (Infections and infestations) | 5 | 4
Gangrene (Infections and infestations) | 4 | 4
Lower respiratory tract infection (Infections and infestations) | 5 | 3
Abscess limb (Infections and infestations) | 6 | 1
Pyelonephritis (Infections and infestations) | 2 | 5
Diverticulitis (Infections and infestations) | 5 | 1
Erysipelas (Infections and infestations) | 3 | 3
Osteomyelitis (Infections and infestations) | 1 | 5
Cystitis (Infections and infestations) | 4 | 1
Localised infection (Infections and infestations) | 2 | 3
Pyelonephritis acute (Infections and infestations) | 4 | 1
Appendicitis (Infections and infestations) | 3 | 1
Bacteraemia (Infections and infestations) | 2 | 2
Bronchopneumonia (Infections and infestations) | 3 | 1
Endocarditis (Infections and infestations) | 2 | 2
Lobar pneumonia (Infections and infestations) | 3 | 1
Subcutaneous abscess (Infections and infestations) | 2 | 2
Wound infection (Infections and infestations) | 4 | 0
Arthritis bacterial (Infections and infestations) | 1 | 2
Gastroenteritis viral (Infections and infestations) | 2 | 1
Herpes zoster (Infections and infestations) | 2 | 1
Respiratory tract infection (Infections and infestations) | 2 | 1
Urosepsis (Infections and infestations) | 2 | 1
Viral infection (Infections and infestations) | 1 | 2
Appendicitis perforated (Infections and infestations) | 1 | 1
Atypical pneumonia (Infections and infestations) | 0 | 2
Carbuncle (Infections and infestations) | 0 | 2
Diarrhoea infectious (Infections and infestations) | 0 | 2
Intestinal gangrene (Infections and infestations) | 1 | 1
Mediastinitis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Wound infection staphylococcal (Infections and infestations) | 0 | 2
Abdominal sepsis (Infections and infestations) | 1 | 0
Abdominal wall infection (Infections and infestations) | 1 | 0
Acinetobacter bacteraemia (Infections and infestations) | 0 | 1
Acute hepatitis B (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Bacterial diarrhoea (Infections and infestations) | 0 | 1
Bacterial pyelonephritis (Infections and infestations) | 0 | 1
Biliary tract infection (Infections and infestations) | 1 | 0
Breast abscess (Infections and infestations) | 1 | 0
Cystitis escherichia (Infections and infestations) | 1 | 0
Dacryocanaliculitis (Infections and infestations) | 0 | 1
Dengue fever (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 1
Diabetic gangrene (Infections and infestations) | 0 | 1
Endocarditis bacterial (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Extradural abscess (Infections and infestations) | 0 | 1
Gas gangrene (Infections and infestations) | 1 | 0
Gastritis viral (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1
Genital infection (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0
HIV infection (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0
Incision site infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0
Korean haemorrhagic fever (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Malaria (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Meningitis viral (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 1
Osteomyelitis acute (Infections and infestations) | 0 | 1
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Periodontitis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pleural infection bacterial (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1
Post procedural cellulitis (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Scrotal abscess (Infections and infestations) | 0 | 1
Scrub typhus (Infections and infestations) | 0 | 1
Serratia infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Thrombophlebitis septic (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1
Urethritis (Infections and infestations) | 0 | 1
Viraemia (Infections and infestations) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 25 | 15
Ischaemic stroke (Nervous system disorders) | 7 | 15
Syncope (Nervous system disorders) | 9 | 9
Transient ischaemic attack (Nervous system disorders) | 7 | 5
Convulsion (Nervous system disorders) | 2 | 7
Carotid artery stenosis (Nervous system disorders) | 5 | 3
Cerebral infarction (Nervous system disorders) | 4 | 4
Epilepsy (Nervous system disorders) | 3 | 2
Haemorrhagic stroke (Nervous system disorders) | 4 | 0
Presyncope (Nervous system disorders) | 2 | 2
Sciatica (Nervous system disorders) | 2 | 2
Carpal tunnel syndrome (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 3 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 2 | 1
Lacunar infarction (Nervous system disorders) | 2 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 2
Carotid artery disease (Nervous system disorders) | 0 | 2
Cauda equina syndrome (Nervous system disorders) | 1 | 1
Cerebrovascular disorder (Nervous system disorders) | 2 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 1
Coma (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 0
Hemiparesis (Nervous system disorders) | 1 | 1
Hypoglycaemic seizure (Nervous system disorders) | 0 | 2
Migraine (Nervous system disorders) | 0 | 2
Neuralgia (Nervous system disorders) | 1 | 1
Neuritis cranial (Nervous system disorders) | 2 | 0
Polyneuropathy (Nervous system disorders) | 2 | 0
Spinal claudication (Nervous system disorders) | 1 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 2
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Brain hypoxia (Nervous system disorders) | 1 | 0
Brain stem haemorrhage (Nervous system disorders) | 0 | 1
Brain stem stroke (Nervous system disorders) | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Carotid sinus syndrome (Nervous system disorders) | 1 | 0
Central pain syndrome (Nervous system disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebral arteriosclerosis (Nervous system disorders) | 1 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0
Diabetic ketoacidotic hyperglycaemic coma (Nervous system disorders) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0
Petit mal epilepsy (Nervous system disorders) | 0 | 1
Senile dementia (Nervous system disorders) | 1 | 0
Thrombotic cerebral infarction (Nervous system disorders) | 0 | 1
VIth nerve paralysis (Nervous system disorders) | 1 | 0
Vascular dementia (Nervous system disorders) | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 36 | 43
Renal failure (Renal and urinary disorders) | 13 | 12
Renal failure chronic (Renal and urinary disorders) | 13 | 9
Renal impairment (Renal and urinary disorders) | 7 | 8
Haematuria (Renal and urinary disorders) | 2 | 5
Nephrolithiasis (Renal and urinary disorders) | 2 | 4
Urinary retention (Renal and urinary disorders) | 0 | 6
Calculus ureteric (Renal and urinary disorders) | 3 | 2
Azotaemia (Renal and urinary disorders) | 3 | 1
Renal colic (Renal and urinary disorders) | 2 | 2
Calculus urinary (Renal and urinary disorders) | 2 | 1
Diabetic nephropathy (Renal and urinary disorders) | 2 | 1
Acute prerenal failure (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Nephropathy (Renal and urinary disorders) | 1 | 1
Prerenal failure (Renal and urinary disorders) | 0 | 2
Renal artery stenosis (Renal and urinary disorders) | 2 | 0
Renal tubular necrosis (Renal and urinary disorders) | 2 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Incontinence (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 1
Renal embolism (Renal and urinary disorders) | 1 | 0
Renal injury (Renal and urinary disorders) | 0 | 1
Renal mass (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 15 | 24
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 19 | 13
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 15 | 13
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 9
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 54 | 40
Chest pain (General disorders) | 9 | 8
Sudden cardiac death (General disorders) | 8 | 8
Sudden death (General disorders) | 7 | 6
Death (General disorders) | 6 | 6
Pyrexia (General disorders) | 3 | 3
Multi-organ failure (General disorders) | 2 | 3
Chest discomfort (General disorders) | 3 | 1
Device occlusion (General disorders) | 2 | 2
Oedema peripheral (General disorders) | 1 | 3
Asthenia (General disorders) | 3 | 0
Adverse drug reaction (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 0 | 2
Cardiac death (General disorders) | 1 | 0
Device battery issue (General disorders) | 1 | 0
Device dislocation (General disorders) | 0 | 1
Device failure (General disorders) | 1 | 0
Hyperpyrexia (General disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 0
Implant site pain (General disorders) | 1 | 0
Necrobiosis (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Pseudoangina (General disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 10 | 9
Diarrhoea (Gastrointestinal disorders) | 8 | 8
Gastritis (Gastrointestinal disorders) | 7 | 3
Pancreatitis (Gastrointestinal disorders) | 4 | 6
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 6
Abdominal pain (Gastrointestinal disorders) | 3 | 6
Gastritis erosive (Gastrointestinal disorders) | 4 | 2
Pancreatitis acute (Gastrointestinal disorders) | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 2
Gastric ulcer (Gastrointestinal disorders) | 3 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 4
Haemorrhoids (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 3 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 2
Duodenal ulcer (Gastrointestinal disorders) | 2 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 3
Inguinal hernia (Gastrointestinal disorders) | 1 | 2
Oesophagitis (Gastrointestinal disorders) | 1 | 2
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 2
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 3
Peptic ulcer (Gastrointestinal disorders) | 2 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Erosive duodenitis (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hernial eventration (Gastrointestinal disorders) | 1 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Intestinal angina (Gastrointestinal disorders) | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Lip haematoma (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1
Pancreatic enlargement (Gastrointestinal disorders) | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Peritonitis sclerosing (Gastrointestinal disorders) | 0 | 1
Retroperitoneal fibrosis (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 17 | 19
Fall (Injury, poisoning and procedural complications) | 6 | 3
Femur fracture (Injury, poisoning and procedural complications) | 8 | 1
Laceration (Injury, poisoning and procedural complications) | 3 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 2
Arterial restenosis (Injury, poisoning and procedural complications) | 0 | 3
Foot fracture (Injury, poisoning and procedural complications) | 2 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 2
Rib fracture (Injury, poisoning and procedural complications) | 3 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 3
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 3 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 2 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2
Overdose (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 2
Pubis fracture (Injury, poisoning and procedural complications) | 2 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 2 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Accident (Injury, poisoning and procedural complications) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Coronary artery reocclusion (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Eyeball rupture (Injury, poisoning and procedural complications) | 1 | 0
Fat embolism (Injury, poisoning and procedural complications) | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Human bite (Injury, poisoning and procedural complications) | 1 | 0
Inflammation of wound (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Open fracture (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 | 0
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Repetitive strain injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Tobacco poisoning (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 1 | 0
Hypertension (Vascular disorders) | 16 | 8
Peripheral arterial occlusive disease (Vascular disorders) | 9 | 9
Hypertensive crisis (Vascular disorders) | 10 | 5
Hypotension (Vascular disorders) | 7 | 6
Peripheral artery stenosis (Vascular disorders) | 1 | 6
Peripheral vascular disorder (Vascular disorders) | 4 | 3
Deep vein thrombosis (Vascular disorders) | 2 | 3
Hypertensive emergency (Vascular disorders) | 2 | 3
Aortic stenosis (Vascular disorders) | 1 | 3
Malignant hypertension (Vascular disorders) | 2 | 2
Peripheral ischaemia (Vascular disorders) | 2 | 2
Hypovolaemic shock (Vascular disorders) | 3 | 0
Intermittent claudication (Vascular disorders) | 0 | 3
Orthostatic hypotension (Vascular disorders) | 0 | 3
Arterial occlusive disease (Vascular disorders) | 2 | 0
Circulatory collapse (Vascular disorders) | 2 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 1
Iliac artery occlusion (Vascular disorders) | 1 | 1
Accelerated hypertension (Vascular disorders) | 1 | 0
Angiodysplasia (Vascular disorders) | 1 | 0
Angiopathy (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Aortic occlusion (Vascular disorders) | 1 | 0
Aortic thrombosis (Vascular disorders) | 0 | 1
Arterial insufficiency (Vascular disorders) | 0 | 1
Arterial stenosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Arteriovenous fistula (Vascular disorders) | 1 | 0
Femoral artery embolism (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1
Subclavian artery stenosis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Venous insufficiency (Vascular disorders) | 0 | 1
Venous occlusion (Vascular disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 16 | 18
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 14 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 11 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 5
Gout (Metabolism and nutrition disorders) | 4 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 5
Dehydration (Metabolism and nutrition disorders) | 4 | 1
Fluid overload (Metabolism and nutrition disorders) | 2 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 1
Diabetes complicating pregnancy (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperosmolar state (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 14 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Signet-ring cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 9 | 7
Cholecystitis (Hepatobiliary disorders) | 2 | 5
Cholecystitis acute (Hepatobiliary disorders) | 2 | 4
Cholecystitis chronic (Hepatobiliary disorders) | 3 | 0
Bile duct stone (Hepatobiliary disorders) | 2 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 2
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Post cholecystectomy syndrome (Hepatobiliary disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 17 | 16
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Haemoglobin decreased (Investigations) | 3 | 0
Lipase increased (Investigations) | 2 | 1
Amylase increased (Investigations) | 0 | 2
Blood glucose increased (Investigations) | 2 | 0
Cardiac enzymes increased (Investigations) | 2 | 0
Hepatic enzyme increased (Investigations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 1 | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Heart rate irregular (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Pancreatic enzymes increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 4 | 7
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 4
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Dry gangrene (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Cataract (Eye disorders) | 6 | 5
Diabetic retinopathy (Eye disorders) | 1 | 1
Vitreous haemorrhage (Eye disorders) | 2 | 0
Amaurosis (Eye disorders) | 1 | 0
Cataract subcapsular (Eye disorders) | 0 | 1
Dacryostenosis acquired (Eye disorders) | 0 | 1
Open angle glaucoma (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Retinopathy (Eye disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 2
Anxiety disorder (Psychiatric disorders) | 1 | 1
Completed suicide (Psychiatric disorders) | 2 | 0
Stress (Psychiatric disorders) | 1 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Agoraphobia (Psychiatric disorders) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 1
Schizophrenia, paranoid type (Psychiatric disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 6 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 1
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Prostatism (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Scrotal mass (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 3
Vertigo positional (Ear and labyrinth disorders) | 2 | 3
Anaphylactic reaction (Immune system disorders) | 3 | 1
Congenital megaureter (Congenital, familial and genetic disorders) | 0 | 1
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 | 0
Goitre (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hospitalisation (Surgical and medical procedures) | 1 | 0
Implantable defibrillator insertion (Surgical and medical procedures) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2679) | Alogliptin (N=2701)
Anaemia (Blood and lymphatic system disorders) | 96 | 130
Angina pectoris (Cardiac disorders) | 133 | 122
Diarrhoea (Gastrointestinal disorders) | 99 | 122
Constipation (Gastrointestinal disorders) | 66 | 70
Nausea (Gastrointestinal disorders) | 53 | 56
Oedema peripheral (General disorders) | 104 | 101
Nasopharyngitis (Infections and infestations) | 120 | 112
Urinary tract infection (Infections and infestations) | 94 | 102
Upper respiratory tract infection (Infections and infestations) | 85 | 79
Bronchitis (Infections and infestations) | 68 | 81
Influenza (Infections and infestations) | 54 | 64
Blood creatine phosphokinase increased (Investigations) | 116 | 140
Glomerular filtration rate decreased (Investigations) | 116 | 132
Lipase increased (Investigations) | 83 | 81
Blood creatinine increased (Investigations) | 72 | 91
Creatinine renal clearance decreased (Investigations) | 47 | 59
Hypoglycaemia (Metabolism and nutrition disorders) | 159 | 167
Hyperglycaemia (Metabolism and nutrition disorders) | 99 | 94
Hyperkalaemia (Metabolism and nutrition disorders) | 70 | 81
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 71 | 55
Diabetes mellitus (Metabolism and nutrition disorders) | 70 | 52
Dyslipidaemia (Metabolism and nutrition disorders) | 49 | 56
Back pain (Musculoskeletal and connective tissue disorders) | 84 | 79
Arthralgia (Musculoskeletal and connective tissue disorders) | 64 | 68
Pain in extremity (Musculoskeletal and connective tissue disorders) | 60 | 54
Dizziness (Nervous system disorders) | 68 | 81
Headache (Nervous system disorders) | 72 | 69
Renal impairment (Renal and urinary disorders) | 174 | 203
Proteinuria (Renal and urinary disorders) | 107 | 103
Diabetic nephropathy (Renal and urinary disorders) | 68 | 62
Cough (Respiratory, thoracic and mediastinal disorders) | 99 | 98
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 74 | 70
Hypertension (Vascular disorders) | 198 | 193

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.